CLINICAL TRIAL: NCT03401580
Title: Clinical Trial to Compare the Efficacy and Safety of Fixed-doses of VIENA II in Participants With Hypertension and Dyslipidemia
Brief Title: Efficacy of Fixed-doses of Antihypertensive and Statin Drugs
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0317
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Hypertension; Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Viena II - 160/10 (Experimental): Fixed-dose, 160mg +10 mg, orally, once daily.
  Interventions: Drug: Viena II 160/10
- Viena II - 190/10 (Experimental): Fixed-dose, 190mg + 10 mg, orally, once daily.
  Interventions: Drug: Viena II 190/10
- Viena II - 160/12 (Experimental): Fixed-dose, 160mg + 12 mg, orally, once daily.
  Interventions: Drug: Viena II 160/12
- Viena II - 190/12 (Experimental): Fixed-dose, 190mg + 12 mg, orally, once daily.
  Interventions: Drug: Viena II 190/12

INTERVENTIONS:
Drug: Viena II 160/10 — once daily
  Other Names: Viena II fixed dose
  Arms: Viena II - 160/10
Drug: Viena II 190/10 — once daily
  Other Names: Viena II fixed dose
  Arms: Viena II - 190/10
Drug: Viena II 160/12 — once daily
  Other Names: Viena II fixed dose
  Arms: Viena II - 160/12
Drug: Viena II 190/12 — once daily
  Other Names: Viena II fixed dose
  Arms: Viena II - 190/12

SUMMARY:
The purpose of this study is to evaluate the efficacy of different fixed-dose combination of Viena II in treatment of hypertension and dyslipidemia.

DETAILED DESCRIPTION:
* Fase II, national, multicenter, randomized, double-blind.
* Maximal duration: 8 weeks;
* 04 visits;
* Safety and efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes aged between 18 and 65 years;
* Participants diagnosed with uncontrolled hypertension (stage 1), according VII Brazilian Guideline of Hypertension;
* Participants diagnosed with dyslipidemia, according to the V Brazilian Guidelines on Dyslipidemia and Prevention of Atherosclerosis;
* Signed consent.

Exclusion Criteria:

* Participants with a previous diagnosis of familial hypercholesterolemia (homozygous);
* Concomitant use of angiotensin II receptor blocker (ARB) or inhibitor of angiotensin converting enzyme (ACE);
* Participants with total cholesterol (TC) above 500 mg / dL or triglyceride (TG) above 500 mg / dL;
* Participants with hypertension (stage 2 or 3) according VII Brazilian Guideline of Hypertension;
* History of congestive heart failure (CHF) functional class III or IV (NYHA);;
* Any clinical, laboratory and electrocardiographic that, in the judgment of the investigator, may interfere with the safety of research participants;
* Creatine phosphokinase (CPK) levels above the established laboratory normal range;
* Transaminases (ALT and ASL) serum above 2 times the established laboratory normal range;
* Body mass index (BMI) ≥35 kg / m²;
* Immunocompromised participants (eg.: malignancies, patients with Acquired Immunodeficiency Syndrome etc);
* Chronic use of drugs that may interact with the drugs of the study;
* History hypersensitivity to the active ingredients used in the study;
* Pregnancy or risk of pregnancy and lactating patients;
* History of alcohol abuse or illicit drug use;
* Participation in clinical trial in the year prior to this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Reduction of systemic blood pressure measured between the first visit and last visit | 8 weeks
Percentage of reduction of LDL-c between the first visit and the last visit. | 8 weeks

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study | 8 weeks